CLINICAL TRIAL: NCT03275129
Title: Pushing the Envelope: Perioperative Cardiorespiratory US for Hip Fractures Procedure
Brief Title: Ultrasound Assessment of Heart and Lungs for Hip Fracture Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Jason Chui, Associate Professor, Anesthesiologist, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: US Hip Fracture
Record Dates: First submitted 2017-08-24; First posted 2017-09-07 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Hip Fractures
Keywords: ultrasound assessment
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Intervention Model Description: Patients over the age of 18 who arrive to the hospital requiring surgery for hip fracture repair.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultrasound assessment of heart and lungs (Experimental): Patients (over the age of 18) who will be undergoing surgery for hip fracture repair. These patients will receive an ultrasound of the heart and lungs to determine whether or not information gained from this ultrasound assessment is significant enough to influence their anesthetic care plan.
  Interventions: Diagnostic Test: Ultrasound assessment of heart and lungs

INTERVENTIONS:
Diagnostic Test: Ultrasound assessment of heart and lungs — Patients will receive an ultrasound assessment of their heart and lungs.

SUMMARY:
The investigators would like to investigate whether performing ultrasound assessments in patients undergoing surgery for hip fractures is able to identify previously undiagnosed heart or lung conditions. The investigators would like to determine whether information provided by this ultrasound assessment is significant enough to alter the anesthetic management plan of these patients. This study has the potential to demonstrate that ultrasound could be used as a diagnostic bedside tool in the perioperative period, possibly altering standard of care for this patient population.

DETAILED DESCRIPTION:
Ultrasound (US) guidance plays an important role in many commonly performed perioperative anesthetic procedures, including central venous catheter (CVC) insertion and regional nerve blocks[1]. The benefits of US guidance in improving patient safety and procedural efficacy have been widely recognized; studies have shown that US guidance reduced the failure rates and the number of attempts required for needle insertion[1, 2]. Multiple national clinical practice guidelines, including those issued by the National Institute for Health and Care Excellence (NICE) in the UK, and the Canadian Anesthesiologists' Society[3, 4], have recommended the routine uses of US guidance for performing invasive anesthetic procedures. The NICE guidelines stated that "US guidance should be used in most clinical circumstances where CVC insertion is necessary and that all those involved in placing CVCs using US guidance should undertake appropriate training to achieve competence[3]." Despite these recommendations, the routine use of US guidance has not been fully adopted by anesthesiologists in South Western Ontario in the past. Matava et al. conducted a survey in 2011 across Ontario and found that only 60% of anesthesiologists at academic hospitals and 33% at community hospitals use US guidance routinely for CVC insertion[5]. In addition, 56% and 31% of academic and community hospital practitioners (respectively) use US guidance routinely for performing regional nerve block[5]. Lack of training and perceived need were identified as the major reasons why they did not routinely use US guidance, reflecting a knowledge gap and deficit in training opportunity in our local region. The interests of using US to provide clinical information in guiding patient management have been demonstrating increasing parallels with the wide availability of US for central line insertion in various settings. Specifically, ultrasound examinations have been developed for emergency medicine (FAST protocol) and intensive care for managing trauma and hemodynamically unstable patients[6]. The same development and application of US has also been true in anesthesia, where the use of Transesophageal echocardiogram has been the standard of care for cardiac surgical procedures for over a decade. The utility of ultrasound for non-cardiac surgery is only just beginning to be explored for perioperative patients, especially for emergency surgery or cases of unexplained hypotension, hemodynamic instability or cardiac arrest. In the past few years, point of care assessment of the heart and lungs with US has become more frequent among anesthesiologists. It was suggested that the uses of US in emergency situations frequently changed the patients' bedside management[7]. The uses of US can also assess volume status and predict hypotension after anesthesia induction. The existing evidence suggests US assessment can lead to more accurate preoperative assessments; however, there is lack of evidence that illustrates how US assessment specifically impacts anesthetic management and patient/procedural outcomes. This information is fundamental to further expand the indications of US applications from purely a procedural guidance tool to a point-of-care diagnostic tool. In Canada, there are approximately 40,000 cases of hip fractures per year[8]. Our institute, the London Health Sciences Centre, in London, Ontario, sees approximately 400 patients a year who have experienced hip fractures and require surgery for treatment. These patients are generally elderly, making this population likely to present with additional comorbidities. Despite the multiple Anesthesia practice guidelines that recommend using US for variety of procedures[3, 4], it is not standard of practice to be used as a preoperative assessment tool for these patients undergoing surgery for hip fractures. Especially considering the advanced age of these patients and potential for underlying comorbidities, using US to assess these patients for cardiac and lung conditions during the perioperative period has the potential to alter their anesthetic management plan if previously undiagnosed conditions are discovered. Introducing the use of point-of-care US assessment for these hip fracture patients has the potential to result in increased patient safety and more favourable patient outcomes. The proposed project involves a prospective cohort study to investigate the utility of US as a clinical assessment tool for patients undergoing hip fracture surgery. In general, patients with hip fractures are elderly with multiple comorbidities, and are at a higher risk for complications. Our current standard of care does not involve the use of US to assess the heart and lung comorbidities of these patients. The use of US has the potential to provide critical information about heart and/or lung diseases that was previously unknown, possibly altering the perioperative management plan and potentially improving care for these patients. Also, careful assessment of the intra vascular volume may help with induction management and Anesthesia technique.The anesthesiologist providing the anesthetic will suggest their anesthesia plan before and after the results of the study will be introduced.

This is a prospective, cohort study. This study will be conducted at the LHSC, London, Ontario. The investigators will include adult patients with a hip fracture scheduled for urgent surgery and exclude patients who have a known heart or lung condition that mandates the appropriate anesthetic plan. Based upon the routine pre-surgical assessments that are performed in accordance with standard of care, the Anesthesiologist will develop and record the plan for anesthetic management for the patient. All patients will receive a preoperative US examination assessment of the heart and lungs (6 basic transthoracic US views ). The US results will be available to the anesthesia and surgical teams, but will only be divulged after a preliminary anesthetic plan is prepared by the anesthesiologist. Following completion of this US assessment, the investigators will ask the Anesthesiologist to re-evaluate their anesthetic plan and document any changes that were made as a result of the US finding and provide feedback about the benefit (or lack thereof) of the information provided by the ultrasound assessment. The primary endpoint of this study is a composite outcome of change in anesthetic technique and choice of monitoring and fluid management. A questionnaire will be distributed to the attending anesthesiologist to record their anesthetic plan pre and post divulgation of US results. The investigators will assess whether the use of perioperative ultrasound provided a significant unknown information that affected the anesthesia plan.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing urgent surgery for hip fractures

Exclusion Criteria:

* under the age of 18 - patients who have a known heart or lung condition that mandates the anesthetic plan

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2018-05-28 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-11 (Actual)

PRIMARY OUTCOMES:
Changes of anesthesiologists' intraoperative management | During surgery
  Changes of anaesthetic management include any changes in postpone of surgery (Y/N), modes of anesthesia (Y/N), uses of EKG (Y/N), arterial line (Y/N), fluid bolus (Y/N), liberal or restrictive fluid management (Y/N), central venous catherization (Y/N), and inotropic uses.

SECONDARY OUTCOMES:
Length of hospital stay | Time to discharge, an average of 2 days
  Patient length of stay will be evaluated
Postoperative complications | Time to discharge, an average of 2 days
  Complications such as cardiac, respiratory and acute kidney injury, blood transfusion will be evaluated for enrolled patients.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Chui, Principal Investigator — University of Western Ontario, Canada
Locations (1):
- LHSC - University Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kline JP. Ultrasound guidance in anesthesia. AANA J. 2011 Jun;79(3):209-17. PMID 21751689
- [Background] Espinet A, Dunning J. Does ultrasound-guided central line insertion reduce complications and time to placement in elective patients undergoing cardiac surgery. Interact Cardiovasc Thorac Surg. 2004 Sep;3(3):523-7. doi: 10.1016/j.icvts.2004.05.006. PMID 17670301
- [Background] Guidance on the Use of Ultrasound Locating Devices for Placing Central Venous Catheters. NICE Guideline, 2002.
- [Background] Merchant R, Chartrand D, Dain S, Dobson G, Kurrek MM, Lagace A, Stacey S, Thiessen B; Canadian Anesthesiologists' Society. Guidelines to the practice of anesthesia--revised edition 2015. Can J Anaesth. 2015 Jan;62(1):54-67. doi: 10.1007/s12630-014-0232-8. PMID 25323121
- [Background] Matava C, Hayes J. A survey of ultrasound use by academic and community anesthesiologists in Ontario. Can J Anaesth. 2011 Oct;58(10):929-35. doi: 10.1007/s12630-011-9555-x. Epub 2011 Jul 12. PMID 21748662
- [Background] Zanobetti M, Coppa A, Nazerian P, Grifoni S, Scorpiniti M, Innocenti F, Conti A, Bigiarini S, Gualtieri S, Casula C, Ticali PF, Pini R. Chest Abdominal-Focused Assessment Sonography for Trauma during the primary survey in the Emergency Department: the CA-FAST protocol. Eur J Trauma Emerg Surg. 2018 Dec;44(6):805-810. doi: 10.1007/s00068-015-0620-y. Epub 2015 Dec 18. PMID 26683569
- [Background] Markin NW, Gmelch BS, Griffee MJ, Holmberg TJ, Morgan DE, Zimmerman JM. A review of 364 perioperative rescue echocardiograms: findings of an anesthesiologist-staffed perioperative echocardiography service. J Cardiothorac Vasc Anesth. 2015 Feb;29(1):82-8. doi: 10.1053/j.jvca.2014.07.004. Epub 2014 Nov 7. PMID 25440641
- [Background] Soong C, Cram P, Chezar K, Tajammal F, Exconde K, Matelski J, Sinha SK, Abrams HB, Fan-Lun C, Fabbruzzo-Cota C, Backstein D, Bell CM. Impact of an Integrated Hip Fracture Inpatient Program on Length of Stay and Costs. J Orthop Trauma. 2016 Dec;30(12):647-652. doi: 10.1097/BOT.0000000000000691. PMID 27875490
- [Derived] Chui J, Hegazy AF, German M, Arango-Ferreira C, Fochesato LA, Lavi R, Bainbridge D. Point-of-care lung and cardiac ultrasound (LUCAS) study in hip fracture patients: a prospective cohort study. Can J Anaesth. 2023 Sep;70(9):1474-1485. doi: 10.1007/s12630-023-02511-5. Epub 2023 Jun 21. PMID 37344745